CLINICAL TRIAL: NCT03787693
Title: Virtual Reality Augmented Gait Adaptation in Stroke Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0291-14-EP
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Stroke
Keywords: hemiparesis; gait; perception; sensory; vision; coordination
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: Chronic stroke survivors will be screened and assigned to either a Symmetric or Asymmetric group based on inter-limb step length and/or step time asymmetry at baseline. Each subject will be randomly assigned to perform a split-belt adaptation protocol in either a VR or a Non-VR environment.
Who Masked: Participant, Investigator
Masking Description: The PI and the subject will not be aware of the group assignment of each subject.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stroke Symmetric Non-VR (No Intervention): In this control arm, stroke survivors who walk symmetrically will walk on a split-belt treadmill in a non-virtual reality environment.
- Stroke Symmetric VR (Experimental): In this experimental arm, stroke survivors who walk symmetrically will walk on a split-belt treadmill in a VR - virtual reality environment.
  Interventions: Behavioral: VR - Virtual Reality
- Stroke Asymmetric Non-VR (No Intervention): In this control arm, stroke survivors who walk asymmetrically will walk on a split-belt treadmill in a non-virtual reality environment.
- Stroke Asymmetric VR (Experimental): In this experimental arm, stroke survivors who walk asymmetrically will walk on a split-belt treadmill in a VR - virtual reality environment.
  Interventions: Behavioral: VR - Virtual Reality

INTERVENTIONS:
Behavioral: VR - Virtual Reality — Subjects in the experimental group will perform the split-belt task in a VR environment
  Arms: Stroke Asymmetric VR; Stroke Symmetric VR

SUMMARY:
The major problem in stroke survivors that is being addressed in this research project is walking asymmetry, i.e., difference between the legs during walking (e.g. steps on the more affected side are longer than the other). A potential solution to this problem is using new technology like virtual reality during walking training to make stroke survivors have a better sense of their asymmetry. A second problem that we aim to address in this study is whether asymmetry is accurately felt by the stroke survivors and how we can address it. Our ongoing work on the effects of virtual reality on learning new walking tasks in stroke survivors indicates that virtual reality maybe particularly important for those with walking asymmetry. In this study, we plan to recruit stroke survivors who have such asymmetries during walking and have them learn a new walking task in virtual reality. We will also test the stroke survivors to determine if there is a relationship between how well they learn the new task with their ability to feel asymmetry accurately.

DETAILED DESCRIPTION:
Stroke survivors show a deterioration in bilateral coordination during gait that impacts functional mobility and quality of life. Such deterioration includes spatial (e.g. step length) and temporal (e.g. step time) inter-limb asymmetries during walking (gait asymmetry). While restoration of gait symmetry through adaptive exercise as in split-belt training is an answer, it is compounded by deficits of perception that is common in stroke survivors. One solution to this problem is the use of augmented visual feedback such as virtual reality (VR). Such augmented visual inputs during training can help remove sensory conflicts that commonly exist during gait rehabilitation (e.g. static visual input versus motion perception through proprioceptive input during treadmill walking). The PI's ongoing research investigating the effects of VR on gait adaptation in stroke survivors indicates that the impact of VR is dependent on the subject's baseline gait asymmetry such that the effect of VR is potentially higher in those who have large baseline asymmetries. Therefore, in the current proposal, to determine if this hypothesis is correct, chronic stroke survivors who are above and below a specific asymmetry threshold will be recruited and assessed for the effect of VR on a split-belt treadmill paradigm. In the second aim, the effect of VR on the transfer of split-belt adaptation to a preferred walking trial will be assessed. Since stroke survivors also suffer from major perceptual deficits related to symmetry, in the third aim, the effect of VR on gait adaptation on four groups of stroke survivors will be analyzed those with deficits only in perceiving visual asymmetry, only gait asymmetry, both deficits or neither.

ELIGIBILITY:
Inclusion Criteria:

* adults > 21 years
* diagnosed with supratentorial ischemic or hemorrhagic stroke
* single, unilateral stroke
* stroke incident > 3 months duration.
* ability to stand unsupported without an assistive device
* walk 10m without therapist assistance,
* ability to follow instructions (Folstein Mini-Mental exam score ≥ 24)

Exclusion Criteria:

* recurrent stroke
* hip fracture
* myocardial infarction
* < 20/40 corrected vision
* any condition that can affect walking ability to complete the experiment successfully (e.g. neglect, Parkinson's disease, vestibulopathy, peripheral nerve pathology).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Step-length Symmetry Index | 1 day
  Difference between the length of a step taken by one limb from the other limb
Step-time Symmetry Index | 1 day
  Difference between the time of a step taken by one limb from the other limb

CONTACTS AND LOCATIONS:
Overall Officials: Mukul Mukherjee, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska - Omaha, Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No